CLINICAL TRIAL: NCT04843033
Title: A Phase I, Open-Label Study to Determine Safety, Tolerability, Pharmacokinetics (PK) and Preliminary Efficacy of SH3809 Tablet in Patients With Advanced Solid Tumors in China
Brief Title: A Study to Investigate Safety and Tolerability of SH3809 Tablet in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing Sanhome Pharmaceutical, Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHC024-I-01
Record Dates: First submitted 2021-04-09; First posted 2021-04-13 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Advanced Solid Tumor
Keywords: advanced solid tum; SHP2; EGFR; NSCLC; Colorectal cancer; KRAS G12
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Daily oral administration of SH3809 tablet (Experimental)
  Interventions: Drug: SH3809 tablet

INTERVENTIONS:
Drug: SH3809 tablet — Starting dose 2mg,oral administered once daily. If tolerated subsequent cohorts will test increasing doses (4mg,6mg,8mg,10mg,12mg) of SH3809.

SUMMARY:
The primary objective is to determine the safety and tolerability of SH3809 in subjects with advanced solid tumors. The second objective is to evaluate the PK profile and preliminary efficacy of SH3809 in solid tumors.

DETAILED DESCRIPTION:
This is a phase I, open-label study to assess the safety,tolerability, pharmacokinetics and preliminary efficacy of SH3809 tablet, a small molecule inhibitor of SHP2 receptor , in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 years inclusive;
2. Histologically or cytologically confirmed advanced malignant solid tumors, eligible patients should be either refractory or intolerant to all available therapies known to confer a clinical benefit as determined by the investigator, except for primary hepatic carcinoma;
3. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1;
4. Life expectancy ≥ 3 months;
5. Adequate hematologic, hepatic and renal function;
6. Participant willing to agree to not father a child/become pregnant and comply with effective contraception criteria;
7. Provision of signed and dated, written informed consent prior to any study-specific evaluation.

Exclusion Criteria:

1. Previous treatment with any SHP2 inhibitors;
2. Spinal cord compression, meningeal metastases or brain metastases unless asymptomatic, stable and not requiring steroids for at least 2 weeks prior to start of study treatment;
3. Life-threatening autoimmune disease or autoimmune disorder with long-term steroid treatment;
4. Active infection with hepatitis B virus (HBV), hepatitis C virus (HCV), human immunodeficiency virus (HIV) and treponema pallidum (TP);
5. Patients who have impaired cardiac function or clinically significant cardiac diseases;
6. Active, clinically significant interstitial lung disease or pneumonitis;
7. Females who are pregnant or breastfeeding;
8. Judgment by the investigator that the patient should not participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2021-04-02 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with dose limiting toxicities (DLTs) | Within the first 28 days of consecutive treatment
  Incidence and nature of DLTs in the dose escalation phase
Maximum tolerated dose(MTD) | Within the first 28 days of consecutive treatment

SECONDARY OUTCOMES:
Cmax | 4 weeks
  Highest observed plasma concentration of SH3809
Tmax | 4 weeks]
  Time of highest observed plasma concentration of SH3809
T1/2 | 4 weeks
  Elimination half-life of SH3809
Area Under the Curve (AUC) | 4 weeks
  Area under the plasma concentration time curve of SH3809
Overall Response Rate(ORR) | up to 12 months
  Overall response rate of SH3809 per RECIST v1.1
Progression-free survival(PFS) | up to 12 months
Disease control rates(DCR) | up to 12 months
  Disease control rates of SH3809 per RECIST v1.1
Duration of response(DOR) | up to 12 months
  Duration of response of SH3809 per RECIST v1.1

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China